CLINICAL TRIAL: NCT03972397
Title: Intercostal Nerve Cryoablation for Postoperative Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Anthony L Estrera, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0283
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Pain, Postoperative
Keywords: Cryoablation
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intercostal Nerve Cryoablation plus SOC Pain Control (Experimental): Standard of Care (SOC)
  Interventions: Device: Intercostal Nerve Cryoablation; Drug: Bupivacaine liposomal injectable suspension; Drug: Patient-controlled analgesia (PCA)
- Standard of Care (SOC) Pain Control (Active Comparator)
  Interventions: Drug: Bupivacaine liposomal injectable suspension; Drug: Patient-controlled analgesia (PCA)

INTERVENTIONS:
Device: Intercostal Nerve Cryoablation — Patients will receive intraoperative intercostal nerve cryoablation using CryoICE® CRYO2 cryoablation probes (AtriCure, Inc) to intercostal spaces 4th to 10th in thoracoabdominal aortic repairs and 4th to 8th in descending thoracic aortic repair cases prior to wound closure.
  Other Names: CryoICE® CRYO2 cryoablation probes (AtriCure, Inc)
  Arms: Intercostal Nerve Cryoablation plus SOC Pain Control
Drug: Bupivacaine liposomal injectable suspension — Patients from both groups will receive the same volume of diluted Exparel®, which will be given in four 20ml syringes using 22-gauge needles (266mg of liposomal bupivacaine, equivalent of one 1.3% 20ml vial of EXPAREL, diluted in 50ml of preservative-free normal (0.9%) sterile saline for a total volume of 70ml).
  Other Names: Exparel® (Pacira Pharmacoceuticals)
Drug: Patient-controlled analgesia (PCA) — Patients will have access to the standard PCA (Patient-Controlled Analgesia) offered at the Memorial Hermann Hospital - Texas Medical Center. The PCA drug will be Dilaudid (hydromorphone). Initial dosing will be per the standard hospital protocol of 0.2 mg demand dose, 10-minute lockout, 2 mg per hour max, 0.4 mg rescue dose. Adjustments to the PCA dosing will be made based on clinical needs.

SUMMARY:
The purpose of the study is to assess the efficacy of intercostal nerve cryoablation on the magnitude and duration of postoperative pain control both in patients undergoing thoracoabdominal incisions for the descending or thoracoabdominal aortic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

* Descending/thoracoabdominal incision is planned
* There is reasonable expectation that the patient will be extubated within 48 hours after surgery

Exclusion Criteria:

* The patient has a known allergy to morphine or any opioid
* The patient has a known chronic pain disorder or takes daily opioid medication > 1 month prior to surgery
* The surgeon/anesthesiologist concludes that the period for intubation will be likely be for more than 48 hours after surgery There is anticipated difficulty communicating pain status due to language or other barriers at the investigator discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L Estrera, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.63) | 54.4 (14.75) | 54.85 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 0 | 0 | 0
  Race/Ethnicity: Asian | 0 | 0 | 0
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race/Ethnicity: Black or African American | 2 | 3 | 5
  Race/Ethnicity: White | 6 | 6 | 12
  Race/Ethnicity: Hispanic | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Score on Numeric Pain Scale (NPS)
Description: The NPS measures the intensity of pain. The total score ranges from 0 to 10, with 0 being no pain and 10 the highest pain.
Time Frame: post-operative day 5
Population: Data were not collected for 2 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 1 participant in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 9
score on a scale | 1.5 [0 to 3.25] | 3 [1 to 4]

2. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: The Brief Pain Inventory is a medical questionnaire used to measure pain, developed by the Pain Research Group of the WHO Collaborating Centre for Symptom Evaluation in Cancer Care. The total severity score ranges from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine.
Time Frame: baseline
Population: Data were not collected for 1 participant in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 10 | 9
score on a scale | 3 [0 to 8] | 6 [0 to 6]

3. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: as for outcome 2
Time Frame: post-operative day 3
Population: Data were not collected for 2 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 2 participants in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 8
score on a scale | 5 [.25 to 10] | 6 [3 to 7.75]

4. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: as for outcome 2
Time Frame: post-operative day 4
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 9
score on a scale | 4.25 [.25 to 7.5] | 7 [6 to 8]

5. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: as for outcome 2
Time Frame: post-operative day 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 9
score on a scale | 4.75 [1 to 8] | 7 [3 to 8]

6. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: as for outcome 2
Time Frame: post-operative day 30
Population: Data were not collected for 1 participant in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 1 participant in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 9 | 9
score on a scale | 5 [2 to 7] | 7 [2 to 8]

7. Primary Outcome: Brief Pain Inventory (BPI) - Severity Score
Description: as for outcome 2
Time Frame: post-operative day 180
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 9 | 9
score on a scale | 2 [0 to 5] | 4 [2 to 8]

8. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: The Brief Pain Inventory is a medical questionnaire used to measure pain, developed by the Pain Research Group of the WHO Collaborating Centre for Symptom Evaluation in Cancer Care. The pain interference score indicates how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. The total pain interference score ranges from 0 to 10, with 0 indicating no interference and 10 indicating complete interference.
Time Frame: baseline
Population: Data were not collected for 1 participant in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 10 | 9
score on a scale | 2.3 [0 to 6] | 0.1 [0 to 4]

9. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: as for outcome 8
Time Frame: post-operative day 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 8
score on a scale | 1.8 [0 to 5.1] | 3.2 [.1 to 4.5]

10. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: as for outcome 8
Time Frame: post-operative day 4
Population: Data were not collected for 5 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 2 participants in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 5 | 8
score on a scale | 1.1 [.1 to 4.3] | 2.9 [.2 to 5.2]

11. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: as for outcome 8
Time Frame: post-operative day 5
Population: Data were not collected for 5 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 4 participants in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 5 | 6
score on a scale | .4 [0 to .9] | 4.6 [1.4 to 6.3]

12. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: as for outcome 8
Time Frame: post-operative day 30
Population: Data were not collected for 4 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 6 participants in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 6 | 4
score on a scale | 2.4 [.1 to 5.0] | 0.1 [0 to 1.1]

13. Primary Outcome: Brief Pain Inventory (BPI) - Pain Interference Score
Description: as for outcome 8
Time Frame: post-operative day 180
Population: Data were not collected for 3 participants in the Intercostal Nerve Cryoablation plus SOC Pain Control arm. Data were not collected for 3 participants in the Standard of Care (SOC) Pain Control arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 7 | 7
score on a scale | 0 [0 to 6.6] | 0 [0 to 5.9]

14. Primary Outcome: 5-point Satisfaction Scale
Description: The 5-point satisfaction scale assesses post-surgical analgesia satisfaction. The total score ranges from 1 to 5, with 1 being "very dissatisfied" and 5 being "very satisfied".
Time Frame: post-operative day 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 8
score on a scale | 5 [3.75 to 5] | 3.5 [2.25 to 4.5]

15. Primary Outcome: 5-point Satisfaction Scale
Description: as for outcome 14
Time Frame: post-operative day 4
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 9
score on a scale | 5 [3.5 to 5] | 3 [3 to 4]

16. Primary Outcome: 5-point Satisfaction Scale
Description: as for outcome 14
Time Frame: post-operative day 5
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 8 | 9
score on a scale | 4.5 [4 to 5] | 4 [2 to 4]

17. Primary Outcome: 5-point Satisfaction Scale
Description: as for outcome 14
Time Frame: post-operative day 30
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 6 | 4
score on a scale | 5 [4 to 5] | 4.5 [4 to 5]

18. Primary Outcome: 5-point Satisfaction Scale
Description: as for outcome 14
Time Frame: post-operative day 180
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 7 | 7
score on a scale | 5 [4 to 5] | 5 [4 to 5]

19. Secondary Outcome: Total Amount in mg of Opioid Medication Consumed
Time Frame: third to fifth post-operative days after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants Who Require of Opioids at the Time of Discharge
Time Frame: at the time of discharge (about a week after surgery)
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Number of Participants Who Utilize Patient-controlled Analgesia (PCA)
Time Frame: from the time immediately after surgery to post-operative day 3
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Amount of Patient-controlled Analgesia (PCA) Used
Time Frame: from the time immediately after surgery to post-operative day 3
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Participants Who Attain Physical Therapy Goal That Justifies Discharge From Inpatient Physical Therapy Within 72 Hours
Time Frame: 72 hours after surgery
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Length of Hospital Stay
Time Frame: at the time of discharge (about a week after surgery)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 10 | 10
days | 10.5 [9 to 13] | 8 [6 to 11]

25. Secondary Outcome: Hospital Cost for Patient Care During Hospitalization
Time Frame: at the time of discharge (about a week after surgery)
Population: Data were not collected for this outcome measure.
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: At time of hospital discharge (about a week after surgery)
Arm/Group | Intercostal Nerve Cryoablation Plus SOC Pain Control | Standard of Care (SOC) Pain Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03972397/Prot_SAP_000.pdf